CLINICAL TRIAL: NCT02467530
Title: Effect of a Low AGE Diet on Human Microbiome
Brief Title: Food Preparation Effects on Gut Bacteria in Patients on Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 14-1961
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: end stage renal disease; peritoneal dialysis (PD); advanced glycation end products; Gut Microbiota Inflammation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Glycation End Products, Advanced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AGE diet (Experimental): Dietary intervention consistent of consuming low amounts of (AGEs).
  Interventions: Other: AGE
- Original diet (No Intervention): Patients will continue their original diet.

INTERVENTIONS:
Other: AGE
  Other Names: Advanced Glycation End products
  Arms: AGE diet

SUMMARY:
This is an intervention study of the effects of food preparation on the gut bacteria in patients with end stage renal disease on peritoneal dialysis. This is a dietary intervention consistent of consuming low amounts of advanced glycation end products (AGEs), the products of protein and sugar interaction during food processing and preparation using high direct heat.

DETAILED DESCRIPTION:
Gut microbes can influence numerous aspects of human biology. Alterations in the function and composition of gut microbial flora (gut microbiota) have been linked to different diseases such as obesity, diabetes and inflammation. Advanced Glycation End products (AGEs) are formed via the Maillard reaction, which consists of a complex network of non-enzymatic reactions involving the carbonyl groups of reducing sugars which react with the amino groups of proteins. AGEs are produced in vivo and being consumed. They have been implicated in increased risk of different diseases including atherosclerosis, CAD and kidney diseases. In this study, the investigators are evaluating the effects of consuming a low AGE diet in participants on peritoneal dialysis on the gut bacteria and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patients with ESRD on PD.
* Patients are able to understand and give consent.
* Patients with estimated daily dietary AGE intake > 12 AGE Eq/day (12,000 kiloUnits/day) based on 3-day food records.

Exclusion Criteria:

* Patient on antibiotics in the last three months.
* Liver cirrhosis, and heart failure with EF < 30%.
* The use of chemotherapy, immunosuppressive medications, probiotics, and steroid in the last month.
* Oral iron supplementation in the last month.
* History of small or large intestine resection or small bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Skin AGE level | baseline and 1 month
  Change in AGE levels in the skin at 1 month compared to baseline will be measure using an AGE reader.

SECONDARY OUTCOMES:
Serum AGE level | baseline and 1 month
  Change in serum AGE level at 1 month compared to baseline
Serum IL-2 level | baseline and 1 month
  Change in serum IL-2 level at 1 month compared to baseline
Serum CRP | baseline and 1 month
  Change in serum CRP level at 1 month compared to baseline
Serum IL-10 | baseline and 1 month
  Change in serum IL-10 level at 1 month compared to baseline
Serum creatinine level | baseline and 1 month
  Change in serum creatinine level at 1 month compared to baseline
Serum blood urea nitrogen (BUN) | baseline and 1 month
  Change in serum BUN at 1 month compared to baseline
Serum p-cresol level | baseline and 1 month
  Change in serum p-cresol level at 1 month compared to baseline
Serum indoxyl sulfate | baseline and 1 month
  Change in serum indoxyl sulfate level at 1 month compared to baseline
Serum vitamin D | baseline and 1 month
  Change in serum vitamin D level at 1 month compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Uribarri, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; John C He, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States